CLINICAL TRIAL: NCT05663931
Title: Implementation and Testing of a Diabetes Discharge Intervention to Improve Safety During Transitions of Care
Brief Title: Diabetes Toolkit at Discharge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Amisha Wallia, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00216291
Record Dates: First submitted 2022-11-17; First posted 2022-12-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Dependent Diabetes
Keywords: Insulin; Hospital discharge; Transitions of care
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DM Discharge Toolkit (Experimental): Up to 60 participants will be recruited for the intervention group. Participants will receive the current standard of care DM education for insulin at Northwestern Memorial Hospital and the adjunctive education with the DM Discharge Toolkit.
  Interventions: Other: DM Discharge Toolkit
- Current Standard of Care Discharge DM Training (No Intervention): Up to 60 participants will be recruited for the control group. Participants will receive the current standard of care DM education for insulin use during current discharge care processes at Northwestern Memorial Hospital.

INTERVENTIONS:
Other: DM Discharge Toolkit — The DM Discharge Toolkit is a multi-modal intervention consisting of a 3-D printed DM survival "kit" that stores DM self-care supplies (e.g., glucose meter) and technical skills (e.g., injection) simulation materials (e.g. simulation skin), whose use is integrated with a website (https://mydiabeteskit.com) containing standardized DM "Survival" education content.
  Arms: DM Discharge Toolkit

SUMMARY:
The purpose of this randomized clinical trial is to implement the DM Discharge Toolkit into hospital discharge and assess the effect of the DM Discharge Toolkit on patients newly requiring insulin.

DETAILED DESCRIPTION:
This study is a randomized controlled trial with a parallel group design of up to 120 study participants in a 1:1 ratio to receive either current standard of care discharge DM training (control) or current standard of care discharge DM training and the DM Discharge Toolkit (intervention) before or immediately after being sent home to assume self-DM care with insulin.

ELIGIBILITY:
Inclusion Criteria:

* English speaking patients
* 18 years of age and older
* Expected survival >90 days
* Need for new insulin at time of hospital discharge

Exclusion Criteria:

* Patients with the inability to give informed consent
* Non-English speaking
* Not diagnosed with diabetes
* Not been newly prescribed insulin

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Mean glucose levels | 30 days
  Mean glucose levels based on home glucose meter and outpatient laboratory data post-discharge

SECONDARY OUTCOMES:
Number of hypoglycemic episodes | 14, 30 and 90 days
  Number of glucoses < 70 mg/dl
Number of hyperglycemic episodes | 14, 30 and 90 days
  Number of blood glucose levels >200 mg/dL
Healthcare utilization | 14, 30 and 90 days
  Number of post-discharge contacts with the healthcare system (i.e. phone calls, emergency room visits, re-admissions, outpatient clinician visits).
HbA1c | 90 days
  Hemoglobin A1c blood test
Time in hyperglycemia | 14 days
  Time in hyperglycemia defined as > 200 mg/dl, outcome from continuous glucose monitor placement
Time in hypoglycemia | 14 days
  Time in hyperglycemia defined as < 70 mg/dl, outcome from continuous glucose monitor placement
Mean amplitude of glycemic excursion | 14 days
  MAGE, outcome from continuous glucose monitor placement
Glycemic variability | 14 days
  A continuous glucose monitor will be used to monitor glucose levels from discharge to 14 days post discharge.
Diabetes Symptoms Questionnaire | 14 days, 30 days
  The Diabetes Symptoms Questionnaire consists of 9 questions where patients answer on a scale between 1-5, with higher numbers indicating a greater rate of occurrence.
Summary of Diabetes Self Care Activities | 14 days, 30 days
  The Summary of Diabetes Self Care Activities consists of 7 questions where patients tally the number of days in the past week that they performed various diabetes self care tasks, such as checking blood glucose and taking medications.
Diabetes Distress Scale | 14 days, 30 days
  The Diabetes Distress Scale is a questionnaire with 17 questions where patients answer on a scale between 1-6, with higher numbers indicating higher distress related to diabetes diagnosis.
Hospital Consumer Assessment of Healthcare Providers and Systems | 14 days, 30 days
  Patient satisfaction survey
Partner Diabetes Distress Scale | Baseline, 30 days, 90 days
  The Partner Diabetes Distress Scale is a questionnaire with 21 questions where a spouse or partner of someone with diabetes answers on a scale between 0-4, with higher numbers indicating higher distress related to partner's diabetes diagnosis.
Perceived Stress Scale | Baseline, 30 days, 90 days
  The Perceived Stress Scale is a questionnaire with 10 questions where a patient answers on a scale between 0-4 with higher numbers indicating a greater rate of occurrence.
Infection | 30 and 90 days
  Rate of infection (bacterial, viral, other)

CONTACTS AND LOCATIONS:
Overall Officials: Amisha Wallia, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No